CLINICAL TRIAL: NCT00816868
Title: A Phase II Study of Erlotinib in Combination With Capecitabine as First-line Treatment in Elderly Patients With Stage IIIB/IV Adenocarcinoma Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Phase II Study of TX Regimen as First-line Treatment for Asian Elderly Patients With Advanced Adenocarcinoma of Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-TONG 0807
Record Dates: First submitted 2009-01-02; First posted 2009-01-05 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: stage IIIB/IV adenocarcinoma non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- non-small cell lung cancer (NSCLC) (Experimental): erlotinib in combination with capecitabine as first-line treatment in elderly patients with stage IIIB/IV adenocarcinoma non-small cell lung cancer (NSCLC)
  Interventions: Drug: erlotinib in combination with capecitabine

INTERVENTIONS:
Drug: erlotinib in combination with capecitabine — Erlotinib 150 mg Q.D. orally for 21 days plus Capecitabine 1000 mg/m2 twice daily for 2 weeks followed by 1 week break every 21 days Until PD, unacceptable toxicity or death.
  Other Names: Tavceva; Xeloda

SUMMARY:
Because of the effect in the treatment of NSCLC, the capecitabine and erlotinib may compose to a new regimen for NSCLC. Based on the preclinical observation and the confirmed clinical synergistic anti-tumor activity of combined capecitabine and erlotinib in gemzar refractory advanced pancreatic cancer (APC), the investigators previously conducted a phase II study of erlotinib in combination with capecitabine against NSCLC.

DETAILED DESCRIPTION:
1. BACKGROUND AND RATIONALE 1.1 Background Lung cancer is the leading cause of cancer-related mortality in the world. Non-small-cell lung cancer (NSCLC), the most common type of lung cancer, comprises about 80% of all lung cancer cases, and five-year survival across all stages is about 12%. More than 60% of all NSCLC patients have advanced or metastatic disease that is not suitable for curative resection at diagnosis. Platinum-based chemotherapy remains the cornerstone of treatment for these patients and results in a small but statistically significant improvement in survival compared with supportive care alone.But the regimen is also associated with moderate to severe hematological and non-hematological toxic effects in a majority of patients.

Approximately two-thirds of patients diagnosed with non-small cell lung cancer (NSCLC) are 65 years or older, and nearly 50% are 70 years or older. And greater than 90% of elderly patients experience a grade 3/4 toxicity when treated with a platinum-based doublet..Moreover，a group of patients with the performance status ≥2 is intolerant intravenous chemotherapy. Availability of an effective,less toxic therapy might help extend potentially beneficial treatment to a greater proportion of elderly or patients whose performance status ≥2.

1.2 Rationale 1.2.1 Capecitabine for NSCLC Capecitabine is an oral prodrug of 5-Fu.It is absorbed through the intestine and converted to 5'-deoxy-S-fluorocytidine (5'-DFCR) by carboxylesterase and then to 5'-deoxy-S-fluorouridine (5'-DFUR) by cytidine deaminase, both steps taking place in the liver. Finally,it is converted to the only active metabolite, FU, by thymidine phosphorylase（TP）. This occurs in both tumor and normal tissues; however, the TP is found at higher concentrations in some tumor tissue compared with normal healthy tissue.The expression of this enzymes may influence the effect of the capecitabine. Han et al examined the TP expression in tumor tissue samples from NSCLC patients who enrolled in a previous phase II study of capecitabine/docetaxel chemotherapy and found that the patients with high tumour cell thymidine phosphorylase expression show a better response to capecitabine based chemotherapy .

The thymidylate synthase (TS) is an important target enzyme for antifolate drugs, such as 5-FU、UFT and capecitabine,because it catalyzes an essential step in DNA synthesis. The predictive role of the expression of thymidylate synthase (TS) in tumors treated with antifolate drugs has been extensively reported in NSCLC.In 2006, Nakano et al performed an immunohistochemical study on the clinical significance of TS expression using 151 resected non-small-cell lung cancer (NSCLC) patients postoperatively treated with UFT.They found that the 5-year survival rate of patients with TS-negative tumours was significantly higher than that with TS-positive tumours (P=0.0133).Miyoshi et al reported that the oral administration of UFT after surgery might improve the survival of NSCLC patients when TS levels in tumor tissues are low,with the 5-year survival rates of patients positive and negative for TS were 50.0 and 89.5%(p<0.001).Some research still found that TS expression was significantly higher in squamous cell carcinoma compared with adenocarcinoma when both mRNA levels and protein levels.

Recently，a Phase III Study Comparing Cisplatin Plus Gemcitabine With Cisplatin Plus Pemetrexed in Chemotherapy-Naïve Patients With Advanced-Stage Non-Small- Cell Lung Cancer showed that Overall survival was statistically superior for cisplatin/ pemetrexed versus cisplatin/gemcitabine in patients with adenocarcinoma.The result reminded us that patients with adenocarcinoma were most likely to benefit from antifolate drugs.

In the preclinical study, we examined tumor specimens for TS and TP expression obtained from 171 Chinese NSCLC patients who were operated without any preoperative chemotherapy or radiation at our institute. We categorized Grades 0 and 1 as negative, Grades 2 and 3 as positive for both enzymes. As for TS staining, 14.6% (n = 25) were classified as Grade 0, 28.7% (n = 49) as Grade 1, 32.7% (n = 56) as Grade 2 and 24.0% (n = 41) as Grade 3. And for TP staining, 12.3% (n = 21) were classified as Grade 0, 17.0% (n = 29) as Grade 1, 13.5% (n = 23) as Grade 2 and 57.3% (n =98) as Grade 3. Although the anti-tumor activity of capecitabine has not been well evaluated in NSCLC, the relatively high expression of TP (70.8%) and low expression TS (43.3%) in NSCLC provided a rationale for the use of capecitabine in patients with this tumor.

1.2.2 Erlotinib for NSCLC Erlotinib is a novel small molecule inhibitor of the EGFR tyrosine kinase (TK). It has been approved as monotherapy for the treatment of patients with advanced NSCLC who have progressed following first- and second-line chemotherapy.It is fairly well tolerated and the salient adverse effects are mild to moderate skin rash and diarrhea. And the further study showed that adenocarcinoma histology predicted the better survival.

Recently a trial of erlotinib as first-line therapy in elderly patients has been reported by investigators at the Dana-Farber Cancer Center. In 76 patients over the age of 70, the vast majority with adenocarcinoma histology, the response rate was 12% and a median survival was 11 months.

1.2.3 The synergistic interaction of erlotinib and capecitabine in NSCLC. Giovannetti et al reported that erlotinib significantly reduced TS expression and activity, possibly via E2F-1 reduction, as detected by RT-PCR and western blot, and the combination decreased TS in situ activity in NSCLC cells. Furthermore, Van SS. et al found TS inhibitor (5-FU) increases EGFR phosphorylation which potentially favors EGFR-TKIs activity.Thus, erlotinib and capecitabine may have a strong synergism in NSCLC.

Because of the effect in the treatment of NSCLC, the capecitabine and erlotinib may compose to a new regimen for NSCLC. Based on the preclinical observation and the confirmed clinical synergistic anti-tumor activity of combined capecitabine and erlotinib in gemzar refractory APC, we previously conducted a phase II study of erlotinib in combination with capecitabine against NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological documented stage IIIB (not amenable for radical /loco-regional therapy) or stage IV (metastatic) adenocarcinoma of lung. Sputum cytology alone is excluded.
2. Measurable disease, according to the Response Evaluation Criteria in Solid Tumours (RECIST), the presence of at least one unidimensionally measurable lesion with longest diameter ≥ 20 mm by conventional techniques OR 10 mm by spiral CT scan.
3. Age ≥ 65.
4. Life expectancy of at least 3 months.
5. Never previously treated with radiotherapy, chemotherapy or surgery for malignant disease.
6. Neutrophil count ≥ 1.5 × 109/L or platelets ≥ 75× 109/L or hemoglobin ≥ 10g/dL
7. Adequate hepatic function including prothrombin time ≥70%of the reference, AST/ALT ≤2.5×institutional upper limit of normal (ULN) or ≤5×ULN if liver metastases, alkaline phosphatase ≤5×ULN (or ≤20×ULN if liver metastases),total bilirubin ≤1.5×ULN
8. Male or female. Age ≥ 18 years.
9. Written (signed) informed consent.
10. Able to comply with study and follow-up procedures.

Exclusion Criteria:

1. Patients with prior surgery or thoracic radiotherapy.
2. Patients with prior chemotherapy or other systemic anti-tumour therapy (e.g. monoclonal antibody therapy or EGFR-TKI) .
3. Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or active peptic ulcer disease.
4. Any inflammatory changes of the surface of the eye.
5. Any diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of any study medication (Erlotinib,Capecitabine) or that might affect the interpretation of the results or render the subject at high risk from treatment complications.
6. Pregnant or lactating women.
7. Woman of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential.
8. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.
9. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal or metabolic disease).
10. History of another malignancy within the last 5 years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix.
11. Patient who are at risk (in the investigator's opinion) of transmitting human immunodeficiency virus (HIV) through blood or other body fluids are excluded.
12. Patients who have brain metastasis or spinal cord compression that has not yet been definitively treated with surgery and/or radiation will be excluded; previously diagnosed and treated CNS metastases or spinal cord compression without evidence of stable disease (clinically stable imaging) for at least 2 months will also be excluded.
13. Hypersensitivity to Erlotinib or Capecitabine

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Non-progression rate (CR + PR + SD) at week 12 and 18 | 1 year
  the percentage of patients who got a complete response, partial response and stable disease at week 12 and at week 18

SECONDARY OUTCOMES:
objective response rate (CR + PR) | 2 year
duration of response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Study Chair — Cancer Center of Sun Yat-Sen University (CCSU)
Locations (1):
- Cancer Center of Sun Yat-Sen University (CCSU), Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhao HY, Chen GY, Huang Y, Li XL, Feng JF, Shi MQ, Cheng Y, Ma LX, Zhang YP, Gu CP, Song XQ, Zhou D, Zhang L. Erlotinib plus capecitabine as first-line treatment for older Chinese patients with advanced adenocarcinoma of the lung (C-TONG0807): an open-label, single arm, multicenter phase II study. Medicine (Baltimore). 2015 Jan;94(2):e249. doi: 10.1097/MD.0000000000000249. PMID 25590835